CLINICAL TRIAL: NCT05436223
Title: A Phase Ⅱ Clinical Study Evaluating the Efficacy and Safety of Human CD19 Targeted T Cells Injection (CD19 CAR-T) Therapy for Relapsed and Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Human CD19 Targeted T Cells Injection(CD19 CAR-T) Therapy for Relapsed and Refractory B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-NHL01-Ⅱ
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: B-cell non-Hodgkin's Lymphoma; CD19; CAR-T; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human CD19 Targeted T Cells Injection (Experimental): Single administration：2.0×10^6 CAR+T/kg
  Interventions: Drug: Human CD19Targeted T Cells Injection

INTERVENTIONS:
Drug: Human CD19Targeted T Cells Injection — A single dose of predetermined level CAR-positive T cells will be infused.
  Other Names: CD19 CAR-T

SUMMARY:
A Phase Ⅱ Clinical Study Evaluating the Efficacy and Safety of Human CD19 Targeted T Cells Injection (CD19 CAR-T) Therapy for R/R B-NHL.

Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19 CAR+ T cells.

DETAILED DESCRIPTION:
Subjects with relapsed and refractory B-cell non-Hodgkin's lymphoma would be selected if subjects meet all criteria evaluated by physical exams, blood tests, electrocardiograph, computedtomography （CT）/magnetic resonance Imaging(MRI)/positron emission tomography（PET）, tumor assessments, etc. Subjects would be hospitalized to receive the infusion of CD19 CAR+ T cells after lymphodepleting regimen, with the observation and evaluation of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:Subjects with relapsed/refractory B-cell non-Hodgkin's lymphoma

* Age≥18 years old，gender is not limited;
* Expected survival > 12 weeks;
* ECOG score 0-2;
* B-cell non-Hodgkin's lymphoma confirmed by cytology or histopathology according to the 2016 World Health Organization (WHO) classification and diagnostic criteria, including: diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed filter Alveolar lymphoma (TFL) and high-grade B-cell lymphoma (HGBCL);
* Pathology demonstrated that B-cell non-Hodgkin's lymphoma and who meet one of the following conditions:

  1. Relapsed and refractory B-cell non-Hodgkin's lymphoma, after standard first-line treatment and at least 2 courses of second-line treatment without remission and relapse (the previous use of CD20-targeted drugs and anthracyclines were needed);
  2. Relapse of B-cell non-Hodgkin lymphoma after stem cell transplantation, regardless of previous treatments.
* The venous access required for collection can be established and leukepheresis can be carried according to the judgement of investigators, satisfying hemoglobin≥80g/L, neutrophils ≥1.0×10^9/L, platelets ≥75×10^9 / L;
* According to the Lugano 2014 criteria, there should be at least one measurable tumor lesion;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Serum creatinine≤1.5×ULN or creatinine clearance rate≥50mL/min (GockcroftGault formula);
  2. Cardiac ejection fraction >50%, no clinically significant pericardial effusion detected, no clinically significant pleural effusion detected;
  3. Baseline blood oxygen saturation>92%;
  4. Total bilirubin≤1.5×ULN(Gilbert syndrome≤5×ULN);
  5. ALT and AST≤3×ULN (AST and ALT ≤5×ULN in patients with liver metastases);
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:Any one of the following conditions cannot be selected as a subject：

* Malignant tumors other than diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), and high-grade B-cell lymphoma (HGBCL) within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection and thyroid cancer after radical resection ;
* Subjects with positive Hepatitis B surface antigen(HBsAg) or Hepatitis B core antibody (HBcAb) and positive peripheral blood hepatitis B virus (HBV) DNA titers (higher than the upper limit of the normal range of the investigative site); Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human Immunodeficiency Viral (HIV) antibody positive; syphilis positive;
* Any uncontrolled systemic diseases, including but not limited to active infection (except for localized infection), uncontrolled angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Any other uncontrolled active disease that precludes participation in the trial;
* Any circumstances that the investigator believes will compromise the safety of the subject or interfere with the purpose of the study;
* Pregnant or lactating woman, or planned pregnancy during treatment or within 1 year after treatment, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment (except uncomplicated urinary tract infection or upper respiratory tract infection);
* Subjects who were receiving systemic steroid treatment within 14 days before enrollment and who were judged by the investigator to require long-term use of systemic steroid therapy during treatment (except inhalation or topical use); or subjects who received any systemic anti-tumor therapy ( except for local anti-tumor therapy) ;
* Subjects who have received CAR-T treatment or other gene-modified cell therapy before enrollment;
* Patients with symptoms of central nervous system or brain metastasis or have received treatment for central nervous system or brain metastasis (radiotherapy, surgery or other treatment) within 3 months before enrollment;
* Subjects who have a disease that affects the signing of written informed consent or who are unable to comply with research procedures; or who are unwilling or unable to comply with research requirements;
* Subjects who are considered unsuitable to participate in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-08-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) at 3 months post infusion | 3 months post infusion
  ORR is defined as proportion of subjects who achieved Partial remission(PR) or better at 3 months (D90±7) post infusion as assessed by an independent review committee (IRC) based on Lugano 2014 criteria.

SECONDARY OUTCOMES:
Duration of remission (DOR) after administration | 2 years post infusion
  DOR refers to the time from the first assessment of complete response or partial response to the first assessment of disease progression or death from any cause.
Progression-free Survival (PFS) after administration | 2 years post infusion
  PFS refers to the time from the start of cell infusion to the first assessment of tumor progression or death from any cause.
Overall Survival (OS) after administration | 2 years post infusion
  OS refers to the time from cell infusion to death due to any cause.
Disease control rate (DCR) | 2 years post infusion
  The best overall response is the ratio of partial response(PR) or complete response(CR) or stable disease(SD) patients to the total number of cases.
Safety evaluation | 2 years post infusion
  The occurrence and outcome of adverse events evaluated by physical examination, laboratory examination, electrocardiogram, imaging scan, etc.
Pharmacokinetic (PK) parameters: Maximum CAR level inperipheral blood | 2 years post infusion
  The highest concentration of Human CD19 Targeted T Cells Injection amplified in peripheral blood after infusion (Cmax) .
Pharmacokinetics(PK) parameters: Time to peak CAR level in blood (Tmax) | 2 years post infusion
  The time to reach the highest concentration of Human CD19 Targeted T Cells Injection in peripheral blood after infusion (Tmax) .
Pharmacokinetics(PK) parameters: 28-day Area under the curve of the CAR level in blood(AUC0-28) | 2 years post infusion
  The 28-day area under the curve of Human CD19 Targeted T Cells Injection in peripheral blood after infusion（AUC0-28d）.
Pharmacodynamic (PD) parameters | 2 years post infusion
  The clearance degree of CD19 positive B cells in peripheral blood at respective time point.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, M.D. & Ph.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No